CLINICAL TRIAL: NCT02292329
Title: Cardiovascular Benefits of Acai in Volunteers at Risk of Metabolic Syndrome.
Brief Title: Cardiovascular Benefits of Acai Polyphenols in Volunteers at Risk of Metabolic Syndrome
Acronym: AF1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AF1UReading
Record Dates: First submitted 2014-09-24; First posted 2014-11-17 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Cardiovascular Diseases
Keywords: flow-mediated dilation; Acai polyphenols
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 150g of acai fruit (Active Comparator): 150g of acai fruit in fruit smoothie form
  Interventions: Dietary Supplement: Acai puree, frozen blended it with banana
- Placebo control (Placebo Comparator): The control will be a smoothie-like drink matched for major macro- and micro-nutrients
  Interventions: Dietary Supplement: Control Macronutrient matched

INTERVENTIONS:
Dietary Supplement: Acai puree, frozen blended it with banana — 150g of acai fruit, frozen blended it with banana.
  Arms: 150g of acai fruit
Dietary Supplement: Control Macronutrient matched — Macronutrient matched control in water and also prepared with banana.
  Arms: Placebo control

SUMMARY:
The purpose of this study is to carry out a randomized double blind controlled trial in 30 male subjects to investigate the effect of acai consumption on acute changes in vascular function, and to other cardiovascular markers. As a secondary aim the study will allow us to characterize the absorption and metabolism of acai polyphenols in humans over a 24 hour period.

ELIGIBILITY:
Inclusion Criteria:

* Male, 30-65 aged, BMI 25-35 kg/m2, Cholesterol <8 mmol/l.

Exclusion Criteria:

* Female, BMI <25 or >35 kg/m2, Cholesterol >8mmol l-1, elevated fasting blood sugar > 6.5 mmols l-1 , elevated systolic blood pressure >150 mmHg, history of stroke or heart attack within the previous 12 months, current smoking, taking lipid lowering, blood pressure lowering or anti-blood clotting medication or taking micronutrient supplements.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation | Change from baseline to 2h

SECONDARY OUTCOMES:
plasma polyphenol metabolites | Change from baseline to 24h

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Commane, PhD, Principal Investigator — University of Reading
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Alqurashi RM, Galante LA, Rowland IR, Spencer JP, Commane DM. Consumption of a flavonoid-rich acai meal is associated with acute improvements in vascular function and a reduction in total oxidative status in healthy overweight men. Am J Clin Nutr. 2016 Nov;104(5):1227-1235. doi: 10.3945/ajcn.115.128728. Epub 2016 Sep 28. PMID 27680990